CLINICAL TRIAL: NCT07279896
Title: Evaluation of Smoking and Oxidative Stress-Induced RNA and DNA Damage in Patients With Stage III Periodontitis
Brief Title: Determination of RNA/DNA Damage Associated With Oxidative Stress in Periodontitis Patients
Status: Completed | Type: Observational
Sponsor: Zehra Hasgül (Other)
Responsible Party: Sponsor-Investigator, Zehra Hasgül, Periodontology Specialist (Resident), Ankara University
Organization: Ankara University (Other)
Other Study IDs: ZH-2025-OxidativeStress
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Periodontitis (Stage 3); Smoking
Keywords: Periodontitis; Smoking; Oxidative Stress; 8-OHdG; 8-OHG; Saliva; Biomarkers
MeSH Terms: conditions — Periodontitis; Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Unstimulated whole saliva samples stored at -80°C. Saliva samples may contain cellular material and DNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Periodontitis Smoker: Participants diagnosed with Stage III periodontitis who are current cigarette smokers. No intervention was applied; biological samples (unstimulated saliva) were collected for biomarker analysis.
- Periodontitis Non-Smoker: Participants diagnosed with Stage III periodontitis who do not smoke. No intervention was applied; unstimulated saliva samples were collected for laboratory analysis.
- Healthy Smoker: Periodontally healthy individuals who are current smokers. No treatment or intervention was performed; only saliva samples and periodontal measurements were obtained.
- Healthy Non-Smoker: Periodontally healthy non-smokers. No intervention was provided; participants underwent periodontal evaluation and saliva sample collection.

SUMMARY:
This study looked at whether a type of gum disease called Stage III periodontitis and cigarette smoking are linked to higher levels of "oxidative stress." Oxidative stress can damage DNA and RNA, which are important parts of our cells. Two markers in saliva-8-OHdG (a sign of DNA damage) and 8-OHG (a sign of RNA damage)-were measured to understand this.

Researchers included four groups of adults: smokers with periodontitis, non-smokers with periodontitis, healthy smokers, and healthy non-smokers. All participants had a dental exam, which checked things like gum inflammation, bleeding, and pocket depth. After the exam, an unstimulated saliva sample was collected from each person. The samples were tested in a laboratory using a sensitive method that measures oxidative damage.

The study found that people with periodontitis had higher levels of DNA and RNA damage in their saliva than healthy people. The highest levels were seen in smokers with periodontitis. Even healthy smokers showed higher levels of oxidative stress than healthy non-smokers. In general, worse gum disease was linked to higher levels of oxidative damage.

These results suggest that saliva tests for 8-OHdG and 8-OHG may help identify gum disease in a simple, non-invasive way. The findings also show that smoking adds to the body's oxidative stress, especially when gum disease is present. The study provides new information about how smoking and gum disease together may affect cell health.

DETAILED DESCRIPTION:
Periodontitis is a chronic inflammatory disease that leads to the progressive destruction of the tooth-supporting tissues. Oxidative stress plays a central role in its pathogenesis, as excessive production of reactive oxygen species (ROS) can damage cellular structures, including lipids, proteins, and nucleic acids. Among oxidative stress-related biomarkers, 8-hydroxy-2'-deoxyguanosine (8-OHdG) and 8-hydroxyguanosine (8-OHG) are widely recognized indicators of DNA and RNA damage, respectively. These biomarkers reflect the biochemical consequences of oxidative stress and are increasingly used to evaluate host responses in periodontal disease.

Cigarette smoking is one of the strongest environmental risk factors for periodontitis and is known to enhance oxidative stress through multiple mechanisms. However, the combined effect of smoking and advanced periodontitis on salivary oxidative DNA and RNA damage has not been fully clarified. Assessing both 8-OHdG and 8-OHG simultaneously may provide deeper insight into the molecular pathways linking smoking, inflammation, and periodontal tissue destruction.

This study was designed to evaluate salivary levels of oxidative nucleic acid damage in individuals with Stage III periodontitis who smoke or do not smoke, as well as in periodontally healthy controls. The study also aimed to investigate the relationship between these biomarkers and clinical periodontal measurements. By examining DNA and RNA oxidation together, the study sought to provide a multidimensional understanding of the host oxidative response in periodontitis.

All participants underwent full-mouth periodontal examination performed by a calibrated clinician. Unstimulated saliva samples were collected under standardized morning conditions, processed by centrifugation to remove cellular debris, and stored at -80°C until biochemical analysis. Levels of 8-OHdG and 8-OHG were quantified using a high-sensitivity ELISA method capable of detecting multiple oxidized guanine derivatives.

Biochemical findings demonstrated that oxidative DNA and RNA damage levels were higher in individuals with periodontitis compared to healthy controls, with smokers exhibiting the highest levels overall. Oxidative biomarker levels showed positive correlations with key periodontal parameters, including probing depth, clinical attachment loss, plaque accumulation, gingival inflammation, and bleeding on probing. These results suggest that the inflammatory burden of periodontitis amplifies oxidative stress at the nucleic acid level and that smoking contributes an additional biological load.

In addition to biochemical assessment, buccal mucosa samples were evaluated cytologically using hematoxylin and eosin staining. All specimens showed adequate cellularity, and no significant differences in epithelial dysplasia were observed across study groups. This may be related to the predominance of superficial epithelial cells in the collected samples.

Overall, this study provides an integrated biochemical and cytomorphological assessment of oxidative stress in periodontitis. The findings support the potential use of salivary 8-OHdG and 8-OHG as non-invasive biomarkers for disease monitoring and contribute novel evidence regarding the interaction between smoking, oxidative stress, and periodontal inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 years or older
* Having at least 16 permanent teeth, excluding third molars
* Not using orthodontic appliances
* Not pregnant or breastfeeding
* Systemically healthy individuals with no systemic diseases that could affect periodontal status
* No use of anti-inflammatory or antimicrobial medications within the last 6 months
* No periodontal treatment within the last 12 months

Exclusion Criteria:

* Pregnant or breastfeeding individuals.
* Use of anti-inflammatory or antimicrobial drugs in the past 6 months.
* Use of antioxidant supplements in the past 3 months.
* Periodontal treatment within the past 12 months.
* Diagnosis of psychiatric disorders.
* Any oral infection.
* Fewer than 16 permanent teeth (excluding third molars).
* Alcohol dependence.
* Active infectious diseases (Acute hepatitis, AIDS, tuberculosis), malignancy, or any systemic condition that may affect periodontal tissues.
* Current use of medications known to affect periodontal tissues (phenytoin, cyclosporine A, calcium channel blockers).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consisted of systemically healthy adults aged 18-65 years, including individuals with Stage III periodontitis and periodontally healthy controls. Participants were categorized into four groups based on periodontal status and smoking habits: smokers and non-smokers with Stage III periodontitis, and smokers and non-smokers who were periodontally healthy.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2025-05-05 (Actual); Primary Completion 2025-08-04 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Salivary oxidative DNA and RNA damage (8-OHdG and 8-OHG levels) | Baseline (periodontal examination visit and saliva collection visit, before any periodontal treatment)
  Concentrations of 8-hydroxy-2'-deoxyguanosine (8-OHdG) and 8-hydroxyguanosine (8-OHG) measured in unstimulated whole saliva using a high-sensitivity competitive ELISA kit. Saliva samples are collected at a separate baseline visit within the study period, after full-mouth periodontal examination and before any periodontal therapy. Biomarker levels (ng/mL) were compared across the four study groups and analyzed in relation to clinical periodontal parameters. Higher values indicate greater oxidative nucleic acid damage.

CONTACTS AND LOCATIONS:
Overall Officials: Sivge Kurgan, Principal Investigator — Ankara University, Faculty of Dentistry, Department of Periodontology
Locations (1):
- Ankara University Faculty of Dentistry, Department of Periodontology, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to patient privacy concerns, data protection regulations, and the terms of the local ethics committee approval

REFERENCES:
- [Result] Hendek MK, Erdemir EO, Kisa U, Ozcan G. Effect of initial periodontal therapy on oxidative stress markers in gingival crevicular fluid, saliva, and serum in smokers and non-smokers with chronic periodontitis. J Periodontol. 2015 Feb;86(2):273-82. doi: 10.1902/jop.2014.140338. Epub 2014 Oct 17. PMID 25325515
- [Result] Tonetti MS, Greenwell H, Kornman KS. Staging and grading of periodontitis: Framework and proposal of a new classification and case definition. J Periodontol. 2018 Jun;89 Suppl 1:S159-S172. doi: 10.1002/JPER.18-0006. PMID 29926952
- [Result] Kurgan S, Onder C, Altingoz SM, Bagis N, Uyanik M, Serdar MA, Kantarci A. High sensitivity detection of salivary 8-hydroxy deoxyguanosine levels in patients with chronic periodontitis. J Periodontal Res. 2015 Dec;50(6):766-74. doi: 10.1111/jre.12263. Epub 2015 Feb 7. PMID 25662588